CLINICAL TRIAL: NCT01469468
Title: A Phase 1, Open-Label, Fixed-Sequence Study To Estimate The Effect Of Repeated Dosing Of PF-05175157 On The Pharmacokinetics Of A Single Dose Of Simvastatin In Healthy Adult Subjects
Brief Title: A Study To Estimate The Effect Of Repeated Dosing of PF-05175157 On The Pharmacokinetics Of A Single Dose Of Simvastatin In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B1731012
Record Dates: First submitted 2011-10-29; First posted 2011-11-10 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm, fixed sequence dosing (Experimental)
  Interventions: Drug: Simvastatin; Drug: PF-05175157

INTERVENTIONS:
Drug: Simvastatin — Day 1: Single dose of simvastatin 20 mg Day 8: single dose of simvastatin 20 mg (with PF-05175157)
Drug: PF-05175157 — Days 2-9 inclusive: daily dosing of PF-05175157 200 mg

SUMMARY:
The study is designed to investigate the effect of repeated dosing of PF-05175157 on the pharmacokinetics of a single dose of Simvastatin in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with normal results in all screening examinations.
* Body Mass Index of 17.5 to 35.5 kg/m2

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, ocular, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Known history of intolerance to simvastatin or other statins.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration curve of simvastatin and simvastatin acid | 10 days
Maximum observed plasma concentration of simvastatin and simvastatin acid | 10 days
Time at which maximum plasma concentration of simvastatin and simvastatin acid is observed | 10 days
If the data permit, area under the plasma concentration curve of simvastatin and simvastatin acid extrapolated to infinite time | 10 days
If the data permit, terminal elimination half-life of simvastatin and simvastatin acid | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States